CLINICAL TRIAL: NCT05411185
Title: The Study on Effects of Acute Exposure to High Altitude Hypoxia on Cognitive Function in Lowlanders
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, DongHailong, Principal Investigator, Xijing Hospital
Other Study IDs: KY20222059
Record Dates: First submitted 2022-05-26; First posted 2022-06-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-02

CONDITIONS: Cognition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the plateau group: People travelling from the plains to areas at altitudes of 3800 meters
- the plain group: People staying in the plains throughout the whole test

SUMMARY:
The purpose of this study is to investigate the impact of rapid elevation to 3,800 meters on the cognitive function of low-altitude residents through a plateau field and plain control study, and explore the objective indicators related to the impaired cognitive function.

DETAILED DESCRIPTION:
This study intends to recruit 60 healthy young people residing in plain area to 3000 m. Participants were divided into two groups: the plateau group (N=30) and the plain group (N=30).

Firstly, we collected baseline data one week before the plateau group rushed to the plateau, and then repeated the above data collection at the same time on day 1 (3-5 hours after arrival), day 2, day 3, day 5, and day 7 after entering the plateau. The plain group was studied in the plain according to the same test plan.

Finally, analyze and find out the main types of cognitive impairment, and explore the physiological prediction index, including exploring the characteristics of EEG changes before and after entering the plateau.

ELIGIBILITY:
Inclusion Criteria:

* Lived in plain, never entered the plateau

Exclusion Criteria:

* patients with epilepsy, migraine, brain injury, stroke and other neuropsychiatric diseases;
* central nervous system drugs;
* history of heart or head surgery;
* MMSE score < 25;
* patients suffering from pulmonary heart disease, chronic obstructive pulmonary disease, emphysema, pulmonary embolism and other serious respiratory diseases;
* patients with negative resistance to the study and poor compliance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: According to the inclusion and exclusion criteria, this study intends to recruit 60 subjects from the healthy young and middle-aged people who live in the plain for the first time, such as students for internship in Tibet for the first time, cadres for aid to Tibet for the first time, and tourists for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cognitive impairment after an altitude of 3,800 meters | 7 days
  To assess cognitive function, we used CNS Vital Signs Neurocognitive test. The core CNS Vital Signs "BRIEF-CORE" neurocognitive assessment battery consists of seven subtests: Verbal Memory (VBM), Visual Memory (VIM), Finger Tapping (FTT), Symbol Digit Coding (SDC), Stroop Test (ST), Rat Attention Test (SAT) and the Continuous Performance Test (CPT). Based on the above 7 test results, the quantitative evaluation results of 11 cognitive functions, including complex memory, graphic memory, vocabulary memory, psychomotor speed, motor speed, processing speed, reaction time, cognitive flexibility, executive function, complex attention and simple attention, were generated.
  By comparing the cognitive function at different stages before and after entering the plateau, we will find out the impaired cognitive function.

SECONDARY OUTCOMES:
The changing trend of cognitive function in plateau environment | 7 days
  For the above 12 cognitive functions, the values in plain and plateau were counted respectively, and then make a line chart to observe the change trend of different cognitive function.
Changes of the relative power values of five different EEG band | 7 days
  To collect the EEG data, we used the ZhenTec's 32-conductivity EEG monitoring device. 32 electrodes ( Fp1、Fp2、F3、F4、Fz、FT7、FT8、FC3、FC4、FCz、Cz、TP7、TP8、CP3、CP4、Pz、Oz、C3、C4、P3、P4、O1、O2、 F7、F8、T3、T4、T5、T6) were placed according to the international 10/20 system electrode placement method, and EEG data of the subjects were collected in the quiet state for 20 min. By analyzing the collected EEG data, we can calculate the relative power values of five different EEG band (δ wave, θ wave, α wave, β wave and γ wave) under different leads.
  By comparing the relative power values at different stages before and after entering the plateau, we tried to look for significantly altered EEG signatures, to find its association with the impaired cognitive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eide RP 3rd, Asplund CA. Altitude illness: update on prevention and treatment. Curr Sports Med Rep. 2012 May-Jun;11(3):124-30. doi: 10.1249/JSR.0b013e3182563e7a. PMID 22580489
- [Background] Ciarlone GE, Dean JB. Acute hypercapnic hyperoxia stimulates reactive species production in the caudal solitary complex of rat brain slices but does not induce oxidative stress. Am J Physiol Cell Physiol. 2016 Dec 1;311(6):C1027-C1039. doi: 10.1152/ajpcell.00161.2016. Epub 2016 Oct 12. PMID 27733363
- [Background] Davranche K, Casini L, Arnal PJ, Rupp T, Perrey S, Verges S. Cognitive functions and cerebral oxygenation changes during acute and prolonged hypoxic exposure. Physiol Behav. 2016 Oct 1;164(Pt A):189-97. doi: 10.1016/j.physbeh.2016.06.001. Epub 2016 Jun 2. PMID 27262217
- [Background] Turner CE, Barker-Collo SL, Connell CJ, Gant N. Acute hypoxic gas breathing severely impairs cognition and task learning in humans. Physiol Behav. 2015 Apr 1;142:104-10. doi: 10.1016/j.physbeh.2015.02.006. Epub 2015 Feb 4. PMID 25660759
- [Background] Falla M, Papagno C, Dal Cappello T, Vogele A, Hufner K, Kim J, Weiss EM, Weber B, Palma M, Mrakic-Sposta S, Brugger H, Strapazzon G. A Prospective Evaluation of the Acute Effects of High Altitude on Cognitive and Physiological Functions in Lowlanders. Front Physiol. 2021 Apr 28;12:670278. doi: 10.3389/fphys.2021.670278. eCollection 2021. PMID 33995130